CLINICAL TRIAL: NCT00598442
Title: AFX01-13: A Phase 3, Randomized, Active-controlled, Open-label, Multi-center Study of the Safety and Efficacy of Peginesatide for the Correction of Anemia in Patients With Chronic Renal Failure (CRF) Not on Dialysis and Not on Erythropoiesis Stimulating Agent (ESA) Treatment
Brief Title: Safety and Efficacy of Peginesatide for the Treatment of Anemia in Participants With Chronic Renal Failure Not on Dialysis
Acronym: PEARL 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Affymax (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-13; 2007-004146-32 (EudraCT Number)
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Renal Failure; Chronic Kidney Disease; Anemia
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia | interventions — peginesatide; hematide; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Peginesatide 0.025 mg/kg (Experimental)
  Interventions: Drug: peginesatide
- Peginesatide 0.04 mg/kg (Experimental)
  Interventions: Drug: peginesatide
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: peginesatide — Participants received peginesatide by subcutaneous injection once every 4 weeks. The starting dose was 0.025 milligram per kilogram (mg/kg) and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 grams per deciliter (g/dL).
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide 0.025 mg/kg
Drug: peginesatide — Participants received peginesatide by subcutaneous injection once every 4 weeks. The starting dose was 0.04 mg/kg and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide 0.04 mg/kg
Drug: Darbepoetin alfa — Participants received darbepoetin alfa by subcutaneous injection once every 2 weeks, as prescribed. The starting dose was 0.75 microgram per kilogram (mcg/kg) and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
  Other Names: Aranesp
  Arms: Darbepoetin alfa

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of peginesatide for the treatment of anemia in participants with chronic kidney disease, who are not on dialysis and not on erythropoiesis stimulating agent (ESA) treatment.

DETAILED DESCRIPTION:
Anemia associated with chronic kidney disease is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The presence and severity of anemia are related to the duration and extent of kidney failure. Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function, and increased left ventricular hypertrophy and heart failure.

Erythropoiesis stimulating agents have been established as a treatment for anemia in chronic renal failure subjects, and have improved the management of anemia over alternatives such as transfusion. Peginesatide is a parenteral formulation developed for the treatment of anemia in patients with chronic kidney disease. Peginesatide binds to and activates the human erythropoietin receptor and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Study participants received doses of peginesatide administered once every 4 weeks or darbepoetin alfa administered once every 2 weeks. Total commitment time for this study was a 4 week screening period followed by a minimum of 52 weeks of study treatment. Eligible participants were randomized in equal proportions to two peginesatide treatment regimens and one control, darbepoetin alfa, treatment regimen.

To evaluate the cardiovascular safety of peginesatide, a cardiovascular composite safety endpoint (CSE) was defined for use in prospectively planned analyses which combined cardiovascular safety data from the four Phase 3 peginesatide studies (NCT00598273, NCT00597753, NCT00598442, and NCT00597584). The CSE consisted of six events: death, stroke, myocardial infarction, and serious adverse events of congestive heart failure, unstable angina, and arrhythmia. An independent Event Review Committee (ERC) was used to provide blinded adjudication of potential CSE events.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic renal failure with an estimated glomerular filtration rate < 60 milliliters per minute per 1.73 m^2 and not expected to begin dialysis for at least 12 weeks.
2. Two consecutive hemoglobin values ≥ 8.0 g/dL and < 11.0 g/dL within 4 weeks prior to randomization.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding.
2. Treatment with an ESA in the 12 weeks prior to randomization.
3. Known intolerance to any ESA, parenteral iron supplementation, or pegylated molecule.
4. Prior chronic hemodialysis or chronic peritoneal dialysis treatment.
5. Known bleeding or coagulation disorder.
6. Known hematologic disease or cause of anemia other than renal disease.
7. Poorly controlled hypertension.
8. Evidence of active malignancy within one year prior to randomization
9. A scheduled kidney transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Affymax
Locations (62):
- United States (41):
  - Research Facility, Phoenix, Arizona
  - Research Facility, Fayetteville, Arkansas
  - Research Facility, Fountain Valley, California
  - Research Facility, Fullerton, California
  - Research Facility, Granada Hills, California
  - Research Facility, Los Angeles, California
  - Research Facility, San Diego, California
  - Research Facility, Whittier, California
  - Research Facility, Lauderdale Lakes, Florida
  - Research Facility, Pembroke Pines, Florida
  - Research Facility, Pinecrest, Florida
  - Research Facility, Canton, Georgia
  - Research Facility, Columbus, Georgia
  - Research Facility, Marietta, Georgia
  - Research Facility, Caldwell, Idaho
  - Research Facility, Meridian, Idaho
  - Research Facility, Chicago, Illinois
  - Research Facility, Mishawaka, Indiana
  - Research Facility, Ames, Iowa
  - Research Facility, Baton Rouge, Louisiana
  - Research Facility, Lafayette, Louisiana
  - Research Facility, Rockville, Maryland
  - Research Facility, Springfield, Massachusetts
  - Research Facility, Detroit, Michigan
  - Research Facility, Flint, Michigan
  - Research Facility, Petoskey, Michigan
  - Research Facility, Troy, Michigan
  - Research Facility, Washington, Missouri
  - Research Facility, Flushing, New York
  - Research Facility, Williamsville, New York
  - Research Facility, Asheville, North Carolina
  - Research Facility, Columbus, Ohio
  - Research Facility, Bend, Oregon
  - Research Facility, Arlington, Texas
  - Research Facility, Houston, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Burlington, Vermont
  - Research Facility, Fairfax, Virginia
  - Research Facility, Tacoma, Washington
  - Research Facility, Morgantown, West Virginia
  - Research Facility, Neenah, Wisconsin
- Bulgaria (3):
  - Research Facility, Sofia
  - Research Facility, Varna
  - Research Facility, Veliko Tarnovo
- Czechia (3):
  - Research Facility, Prague
  - Research Facility, Tábor
  - Research Facility, Zdar
- Research Facility, Demmin, Germany
- Hungary (3):
  - Research Facility, Balatonfüred
  - Research Facility, Kistarcsa
  - Research Facility, Szigetvár
- Italy (2):
  - Research Facility, Lecco
  - Research Facility, Pavia
- Poland (4):
  - Research Facility, Bialystok
  - Research Facility, Gdansk
  - Research Facility, Katowice
  - Research Facility, Zamość
- Research Facility, Ponce, Puerto Rico
- Romania (3):
  - Research Facility, Iași
  - Research Facility, Oradea
  - Research Facility, Timișoara
- Research Facility, London, United Kingdom

REFERENCES:
- [Result] Macdougall IC, Provenzano R, Sharma A, Spinowitz BS, Schmidt RJ, Pergola PE, Zabaneh RI, Tong-Starksen S, Mayo MR, Tang H, Polu KR, Duliege AM, Fishbane S; PEARL Study Groups. Peginesatide for anemia in patients with chronic kidney disease not receiving dialysis. N Engl J Med. 2013 Jan 24;368(4):320-32. doi: 10.1056/NEJMoa1203166. PMID 23343062
- [Derived] Fishbane S, Schiller B, Locatelli F, Covic AC, Provenzano R, Wiecek A, Levin NW, Kaplan M, Macdougall IC, Francisco C, Mayo MR, Polu KR, Duliege AM, Besarab A; EMERALD Study Groups. Peginesatide in patients with anemia undergoing hemodialysis. N Engl J Med. 2013 Jan 24;368(4):307-19. doi: 10.1056/NEJMoa1203165. PMID 23343061

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginesatide 0.025 mg/kg: Participants received peginesatide by subcutaneous injection once every 4 weeks. The starting dose was 0.025 milligram per kilogram (mg/kg) and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 grams per deciliter (g/dL).
- Peginesatide 0.04 mg/kg: Participants received peginesatide by subcutaneous injection once every 4 weeks. The starting dose was 0.04 mg/kg and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
Period: Overall Study
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Started | 167 | 163 | 163
Completed | 124 | 124 | 139
Not Completed | 43 | 39 | 24
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Death | 19 | 11 | 11
Not completed — Lost to Follow-up | 4 | 3 | 3
Not completed — Physician Decision | 2 | 1 | 1
Not completed — Withdrawal by Subject | 8 | 16 | 6
Not completed — Noncompliance | 0 | 2 | 1
Not completed — Relocation | 1 | 4 | 0
Not completed — Renal transplant | 0 | 0 | 1
Not completed — Site closed by sponsor | 5 | 2 | 1
Not completed — Started dialysis | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa | Total
Number analyzed (Participants) | 167 | 163 | 163 | 493
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 63 | 57 | 62 | 182
  >=65 years | 104 | 106 | 101 | 311
Age Continuous [Mean (Standard Deviation); unit: years] | 68.1 (12.93) | 68.3 (13.53) | 67.2 (15.03) | 67.9 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 96 | 99 | 288
  Male | 74 | 67 | 64 | 205

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Between Baseline and the Evaluation Period
Description: The baseline hemoglobin value is defined as the mean of three hemoglobin values: the two most recent hemoglobin values taken prior to the day of randomization and the value obtained on the day of randomization. The mean hemoglobin during the Evaluation Period for each participant is calculated as the mean of the available hemoglobin values during Study Weeks 25 through 36.
Time Frame: Baseline and Weeks 25-36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Number analyzed (Participants) | 167 | 163 | 163
g/dL
  Baseline [N=167, 163, 163] | 10.02 (0.626) | 10.03 (0.618) | 10.03 (0.654)
  Evaluation Period [N=151, 145, 150] | 11.55 (0.741) | 11.71 (0.855) | 11.40 (0.728)
  Change from Baseline [N=151, 145, 150] | 1.50 (0.898) | 1.68 (0.962) | 1.35 (1.004)
Statistical Analysis 1: Comparison: Peginesatide 0.025 mg/kg vs Darbepoetin Alfa; The sample size for this study was determined based on a two-group evaluation of non-inferiority in means with a non-inferiority margin (Δ) of -1.0 g/dL (one-sided significance level of 0.0125, or, comparably, a two-sided significance level of 0.025). A sample size of 450 (150 per treatment group) provided power greater than 99% for the evaluation of non-inferiority, assuming an expected treatment difference of 0.0 g/dL and a pooled standard deviation of 1.5 g/dL; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of -1.0 g/dL was used in the primary efficacy assessments. Non-inferiority was established if the lower limit of the two-sided 97.5% CI for the difference between the means of the primary endpoint (peginesatide minus control ESA) was ≥ -1.0 g/dL; ANOVA; The ANOVA cell means model was used to estimate primary efficacy endpoint within the specified cells formed by the combination of treatment and strata; Least Squares Mean Difference = 0.14, 97.5% CI 2-sided [-0.09 to 0.36], Standard Error of Mean 0.101
Statistical Analysis 2: Comparison: Peginesatide 0.04 mg/kg vs Darbepoetin Alfa; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.31, 97.5% CI 2-sided [0.08 to 0.54], Standard Error of Mean 0.102

2. Secondary Outcome: Proportion of Participants Who Received Red Blood Cell (RBC) Transfusions During the Correction and Evaluation Periods
Time Frame: Weeks 0 to 36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Number analyzed (Participants) | 167 | 163 | 163
percentage of participants | 0.114 | 0.104 | 0.049
Statistical Analysis 1: Comparison: Peginesatide 0.025 mg/kg vs Darbepoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 2.28, 95% CI 2-sided [1.04 to 5.01]
Statistical Analysis 2: Comparison: Peginesatide 0.04 mg/kg vs Darbepoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 2.10, 95% CI 2-sided [0.94 to 4.69]

3. Secondary Outcome: Proportion of Participants Achieving Hemoglobin Response During the Correction and Evaluation Periods
Description: A hemoglobin response is defined as a hemoglobin increase of ≥ 1.0 gram per deciliter (g/dL) above baseline and a hemoglobin ≥ 11.0 g/dL without RBC transfusion during the previous 8 weeks.
Time Frame: Weeks 0 to 36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Number analyzed (Participants) | 167 | 163 | 163
percentage of participants | 0.910 | 0.933 | 0.951
Statistical Analysis 1: Comparison: Peginesatide 0.025 mg/kg vs Darbepoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.90 to 1.01]
Statistical Analysis 2: Comparison: Peginesatide 0.04 mg/kg vs Darbepoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.93 to 1.04]

ADVERSE EVENTS:
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 86/167 | 80/163 | 70/163
Other Adverse Events (participants affected / at risk) | 142/167 | 134/163 | 134/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide 0.025 mg/kg (N=167) | Peginesatide 0.04 mg/kg (N=163) | Darbepoetin Alfa (N=163)
Anaemia (Blood and lymphatic system disorders) | 7 | 6 | 4
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 7 | 18 | 12
Acute myocardial infarction (Cardiac disorders) | 5 | 4 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 5 | 4
Cardiac arrest (Cardiac disorders) | 5 | 2 | 3
Myocardial infarction (Cardiac disorders) | 4 | 2 | 4
Bradycardia (Cardiac disorders) | 4 | 5 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 3 | 1
Angina unstable (Cardiac disorders) | 3 | 2 | 0
Cardiac failure (Cardiac disorders) | 2 | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 2 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 5 | 2
Pancreatitis acute (Gastrointestinal disorders) | 2 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastric hypomotility (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0
Uraemic gastropathy (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 4 | 1
Pyrexia (General disorders) | 1 | 1 | 2
Generalised oedema (General disorders) | 1 | 2 | 0
Asthenia (General disorders) | 2 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1
Multi-organ failure (General disorders) | 2 | 0 | 0
Brain death (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 3 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0
Transplant rejection (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 11 | 5
Urinary tract infection (Infections and infestations) | 5 | 5 | 1
Cellulitis (Infections and infestations) | 4 | 2 | 3
Lobar pneumonia (Infections and infestations) | 3 | 2 | 0
Sepsis (Infections and infestations) | 0 | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 2 | 1
Osteomyelitis (Infections and infestations) | 1 | 2 | 1
Bacteraemia (Infections and infestations) | 0 | 2 | 1
Wound infection (Infections and infestations) | 2 | 1 | 0
Gangrene (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile sepsis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0
Diabetic gangrene (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis bacterial (Infections and infestations) | 0 | 1 | 0
Perihepatic abscess (Infections and infestations) | 0 | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia cryptococcal (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 | 0
Coagulation time prolonged (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 6 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Neuroglycopenia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 3
Headache (Nervous system disorders) | 1 | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
Hypoxic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Uraemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 1 | 3
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 11 | 11 | 5
Renal failure chronic (Renal and urinary disorders) | 10 | 6 | 8
Renal failure (Renal and urinary disorders) | 2 | 2 | 1
Azotaemia (Renal and urinary disorders) | 2 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 4
Hypertensive crisis (Vascular disorders) | 3 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 1
Hypertension (Vascular disorders) | 2 | 1 | 1
Aortic aneurysm (Vascular disorders) | 2 | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 2 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0 | 0
Angiopathy (Vascular disorders) | 1 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Cardiovascular insufficiency (Vascular disorders) | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide 0.025 mg/kg (N=167) | Peginesatide 0.04 mg/kg (N=163) | Darbepoetin Alfa (N=163)
Anaemia (Blood and lymphatic system disorders) | 13 | 9 | 4
Hyperparathyroidism (Endocrine disorders) | 8 | 4 | 9
Hyperparathyroidism secondary (Endocrine disorders) | 5 | 9 | 6
Nausea (Gastrointestinal disorders) | 27 | 25 | 27
Diarrhoea (Gastrointestinal disorders) | 22 | 21 | 32
Vomiting (Gastrointestinal disorders) | 17 | 23 | 15
Constipation (Gastrointestinal disorders) | 12 | 16 | 18
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 9 | 5
Abdominal pain (Gastrointestinal disorders) | 9 | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 8 | 6 | 9
Oedema peripheral (General disorders) | 45 | 26 | 34
Fatigue (General disorders) | 15 | 18 | 14
Asthenia (General disorders) | 12 | 8 | 8
Pain (General disorders) | 10 | 2 | 3
Nasopharyngitis (Infections and infestations) | 22 | 19 | 24
Urinary tract infection (Infections and infestations) | 22 | 22 | 22
Upper respiratory tract infection (Infections and infestations) | 12 | 15 | 19
Bronchitis (Infections and infestations) | 5 | 14 | 13
Sinusitis (Infections and infestations) | 5 | 5 | 12
Fall (Injury, poisoning and procedural complications) | 16 | 11 | 10
Contusion (Injury, poisoning and procedural complications) | 13 | 11 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 23 | 24 | 23
Hyperphosphataemia (Metabolism and nutrition disorders) | 16 | 6 | 15
Gout (Metabolism and nutrition disorders) | 11 | 4 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 11 | 6
Iron deficiency (Metabolism and nutrition disorders) | 10 | 4 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 10 | 3 | 8
Anorexia (Metabolism and nutrition disorders) | 9 | 4 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 7 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 16 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 18 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 17 | 17
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 10 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 4 | 14
Dizziness (Nervous system disorders) | 17 | 20 | 20
Headache (Nervous system disorders) | 15 | 15 | 12
Insomnia (Psychiatric disorders) | 13 | 7 | 7
Depression (Psychiatric disorders) | 11 | 7 | 7
Anxiety (Psychiatric disorders) | 10 | 7 | 3
Renal failure chronic (Renal and urinary disorders) | 9 | 4 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 17 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 17 | 16
Hypertension (Vascular disorders) | 32 | 24 | 34
Hypotension (Vascular disorders) | 15 | 13 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the primary safety and efficacy results will include data from all appropriate study sites. Either after the first multicenter publication, or following 36 months after the completion of the study, Investigators are free to publish; such publications may not contain Sponsor Confidential Information and may be subject to Sponsor review 60 days prior to submission for publication.